CLINICAL TRIAL: NCT00384540
Title: Allograft Vasculopathy After Heart Transplantation : Diagnostic Interest of Dobutamine Stress Echocardiography and Brain Natriuretic Peptide Coupling
Brief Title: Cardiac Allograft Vasculopathy and Dobutamine Stress Echocardiography / Brain Natriuretic Peptide Coupling
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 3660
Record Dates: First submitted 2006-10-05; First posted 2006-10-06 (Estimated); Last update posted 2018-07-10 (Actual); Status verified 2017-08

CONDITIONS: Vasculopathy; Allograft
Keywords: -Heart Transplant, Allograft Vasculopathy, Dobutamine Stress Echocardiography, Brain Natriuretic Peptide; Vasculopathy
MeSH Terms: conditions — Vascular Diseases

ARMS (1):
- Cardiovascular events vs Dobutamine stress echocardiography (Other)
  Interventions: Procedure: Dobutamine stress echocardiography, coronarography, brachial arterial echography

INTERVENTIONS:
Procedure: Dobutamine stress echocardiography, coronarography, brachial arterial echography — DSE: cumulative doses of dobutamine (max = 40 µg/kg/min) and atropine (max = 1.5 mg), to reach a maximal heart rate under clinical, electrocardiographic and echocardiographic surveillancesCoronarography: invasive injection into coronary arteries of a radiological product showing a contrast visible on an x-ray. FMD: Flow-mediated dilatation of the brachial artery induced by 5-min forearm arterial occlusion

SUMMARY:
Primary purpose :To early detect cardiac allograft vasculopathy and to identify patients with high risk of cardiac events, by coupling the analysis of the kinetics of the brain natriuretic peptide ( BNP) with that of the left ventricle (LV) during a dobutamine stress echocardiography.

Hypothesis : Plasma BNP elevation and abnormalities of LV kinetic during the ESD, will be associated with the presence of allograft vasculopathy and the arisen of cardiovascular events.

ELIGIBILITY:
Inclusion criteria:

* Heart transplant recipients

Exclusion criteria:

* No respect of inclusion criteria
* Pregnancy
* Severe renal failure (creatinin clearance < or equal to 30 ml/min)
* Dobutamine stress echocardiography contraindication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2006-09 (Actual); Primary Completion 2015-11-22 (Actual); Study Completion 2016-12-20 (Actual)

PRIMARY OUTCOMES:
Cardiovascular events vs Dobutamine stress echocardiography each 2 years | 5 years

SECONDARY OUTCOMES:
Flow mediated humeral dilatation each 2 years | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Samy TALHA, MD, Principal Investigator — Hôpitaux Universitaires de Strasbourg
Locations (1):
- Service de Physiologie et d'Explorations Fonctionnelles, Hôpital Civil, Hôpitaux Universitaires de Strasbourg, Strasbourg, France